CLINICAL TRIAL: NCT03808506
Title: Relationship Between Baseline Burden of Disease and Anti-TNF Drug Trough Levels in Ulcerative Colitis.
Brief Title: Relationship Between Baseline Burden of Disease and TDM in Ulcerative Colitis
Status: Withdrawn | Type: Observational
Why Stopped: no recruitment during COVID pandemic
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Brian Yan, Associate Professor of Medicine, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 113446
Record Dates: First submitted 2019-01-14; First posted 2019-01-17 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Therapeutic drug monitoring; fecal calprotectin; adalimumab; bowel ultrasound
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ulcerative colitis patients: Patients with documented ulcerative colitis who are initiating adalimumab therapy will have baseline bowel ultrasound and fecal calprotectin completed.
  Interventions: Diagnostic Test: Fecal calprotectin

INTERVENTIONS:
Diagnostic Test: Fecal calprotectin — Stool test to look at baseline burden of inflammation

SUMMARY:
Ulcerative colitis (UC) is a chronic inflammatory bowel disease which often follows a relapsing/remitting course. Anti-TNF therapies are proven to be effective in UC and studies indicate that having adequate drug levels correlate with improved patient outcomes. It is unknown, however, if a high burden of disease at baseline impacts drug utilization or loss. In this study, we investigate whether measures of high burden of disease (fecal calprotectin, bowel ultrasound, and colonoscopy) at baseline predicts low drug levels after standard anti-TNF induction therapy.

DETAILED DESCRIPTION:
Biologic therapy has revolutionized the treatment of IBD. Over the past 20 years, a significant amount of research has been done to optimize biologic therapy using therapeutic drug monitoring (TDM). Evidence is accumulating suggesting that insufficient anti-TNF drug levels +/- development of anti-drug antibodies result in lower clinical efficacy, reduced mucosal healing, and loss of response. The pharmacokinetics of anti-TNF drug clearance leading to sub-therapeutic or absent drug levels can vary between and within any given patient. Clearance may be dependent on many factors such as severity of inflammation, total burden of disease, body weight, serum albumin levels, loss of drug through leaking into the stool, and immune mediated pathways with the development of anti-drug antibodies. Standard induction dosing does not take into account the severity and total burden of disease, which may have significant effects on the elimination of circulating drug.

Most data surrounding TDM pertain to maintenance of remission, during a relatively stable state of low burden of disease. Much less is known surrounding active drug levels during or immediately after induction therapy, at which point disease burden is relatively high and fluctuating. Some studies suggest improved response rates in those with higher anti-TNF drug levels during this phase of therapy. A retrospective study by Gibson et al assessed inpatients with acute severe ulcerative colitis and demonstrated reduction in colectomy rates in those who received accelerated and intensified infliximab induction therapy. Although trough levels were not provided in this study, the results suggest that standard induction dosing may be suboptimal in a setting of high burden of disease.

Colonoscopy is considered the gold standard in regards to determining burden of active disease in ulcerative colitis. However, it is invasive, requires endoscopy time, and carries risk. Non-invasive methods to determine the presence and extent of inflammation is of clinical and research interest. Fecal calprotectin (FC) is a promising tool which has now been incorporated into standard clinical care of IBD patients. It is used to monitor disease activity, assess response to therapy, and prognosticate future clinical relapse. Several meta-analyses demonstrate the correlation between FC with endoscopic disease scores in both Crohn's disease (CD) and Ulcerative Colitis (UC) with a pooled sensitivity of 85-92% and specificity of 75-88%.

Bowel Ultrasound (US) is another non-invasive method to assess inflammatory activity in UC, and is used in routine clinical practice. Bowel US correlates to inflammatory activity on colonoscopy and can be used to assess response to therapy and prognosticate future relapse. A benefit of sonography, as compared to colonoscopy and FC, is its ability to identify inflammatory changes deep to the superficial mucosa. This may provide additional information for burden of disease not recognized by other modalities. It is currently unknown if the burden of disease as found on sonography influences drug elimination and the resultant trough levels after induction therapy.

It is unknown if a high burden of disease at baseline impacts drug utilization or loss. In this study, measures of burden of disease (FC, bowel US, and colonoscopy) at baseline will be correlated to drug levels after standard anti-TNF induction therapy. It is hypothesized that a high burden of disease leads to low drug levels after standard induction dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Adult outpatients >=18 y of age with a confirmed diagnosis of ulcerative colitis
2. Patients beginning adalimumab for active disease as clinically indicated according to the treating physician's discretion, either biologic naïve or switching biologic due to failure of prior biologic therapy
3. Have had a colonoscopy or flexible sigmoidoscopy within 12 weeks of study entry
4. Any other concomitant therapies are allowed (including 5'ASA, corticosteroids, azathioprine, and methotrexate).

Exclusion Criteria:

1. Inability to provide informed consent
2. Inability to provide a fecal calprotectin
3. Contraindication to starting anti-TNF therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with documented ulcerative colitis with active inflammation who are starting adalimumab therapy. All other concomittant therapies are allowed.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-06-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Baseline fecal calprotectin concentration | Performed within 4 weeks of starting adalimumab therapy
  Fecal calprotectin concentration at baseline prior to starting adalimumab therapy. Fecal Calprotectin will be used as the primary outcome measure to determine burden of inflammation

SECONDARY OUTCOMES:
Post Induction fecal calprotectin concentration | Performed 6 weeks post induction therapy
  Fecal calprotectin concentration will be re-assessed at week 6 after starting adalimumab therapy
Baseline Mayo Endoscopic Score | Performed within 12 weeks of study entry
  Baseline endoscopic score (as assessed by colonoscopy or flexible sigmoidoscopy) to grade the severity of mucosal inflammation. The Mayo Endoscopic score is a standard, validated, and accepted grading systems which grades inflammation from 0-3.
Baseline bowel ultrasound inflammatory score | Performed within 12 weeks of starting adalimumab therapy
  Baseline severity of inflammation based on sonographic features including bowel wall thickness, depth of mural inflammation, and degree of hypervascularity. Each component will be scored from 0-3 resulting in an ultrasound severity score of 0-9 for the segment assessed. Three segments of the colon (right colon, transverse, left colon) will be assessed and scores combined to give a total inflammatory score.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Yan, H.B Sc, MD, Principal Investigator — Western University
Locations (1):
- London Health Sciences Center, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vande Casteele N, Herfarth H, Katz J, Falck-Ytter Y, Singh S. American Gastroenterological Association Institute Technical Review on the Role of Therapeutic Drug Monitoring in the Management of Inflammatory Bowel Diseases. Gastroenterology. 2017 Sep;153(3):835-857.e6. doi: 10.1053/j.gastro.2017.07.031. Epub 2017 Jul 31. PMID 28774547
- [Background] Mitrev N, Vande Casteele N, Seow CH, Andrews JM, Connor SJ, Moore GT, Barclay M, Begun J, Bryant R, Chan W, Corte C, Ghaly S, Lemberg DA, Kariyawasam V, Lewindon P, Martin J, Mountifield R, Radford-Smith G, Slobodian P, Sparrow M, Toong C, van Langenberg D, Ward MG, Leong RW; IBD Sydney Organisation and the Australian Inflammatory Bowel Diseases Consensus Working Group. Review article: consensus statements on therapeutic drug monitoring of anti-tumour necrosis factor therapy in inflammatory bowel diseases. Aliment Pharmacol Ther. 2017 Dec;46(11-12):1037-1053. doi: 10.1111/apt.14368. Epub 2017 Oct 13. PMID 29027257
- [Background] Steenholdt C, Bendtzen K, Brynskov J, Ainsworth MA. Optimizing Treatment with TNF Inhibitors in Inflammatory Bowel Disease by Monitoring Drug Levels and Antidrug Antibodies. Inflamm Bowel Dis. 2016 Aug;22(8):1999-2015. doi: 10.1097/MIB.0000000000000772. PMID 27135483
- [Background] Maser EA, Villela R, Silverberg MS, Greenberg GR. Association of trough serum infliximab to clinical outcome after scheduled maintenance treatment for Crohn's disease. Clin Gastroenterol Hepatol. 2006 Oct;4(10):1248-54. doi: 10.1016/j.cgh.2006.06.025. Epub 2006 Aug 22. PMID 16931170
- [Background] Paul S, Del Tedesco E, Marotte H, Rinaudo-Gaujous M, Moreau A, Phelip JM, Genin C, Peyrin-Biroulet L, Roblin X. Therapeutic drug monitoring of infliximab and mucosal healing in inflammatory bowel disease: a prospective study. Inflamm Bowel Dis. 2013 Nov;19(12):2568-76. doi: 10.1097/MIB.0b013e3182a77b41. PMID 24013361
- [Background] Ricciuto A, Dhaliwal J, Walters TD, Griffiths AM, Church PC. Clinical Outcomes With Therapeutic Drug Monitoring in Inflammatory Bowel Disease: A Systematic Review With Meta-Analysis. J Crohns Colitis. 2018 Nov 15;12(11):1302-1315. doi: 10.1093/ecco-jcc/jjy109. PMID 30107416
- [Background] Berends SE, Strik AS, Lowenberg M, D'Haens GR, Mathot RAA. Clinical Pharmacokinetic and Pharmacodynamic Considerations in the Treatment of Ulcerative Colitis. Clin Pharmacokinet. 2019 Jan;58(1):15-37. doi: 10.1007/s40262-018-0676-z. PMID 29752633
- [Background] Berends SE, Strik AS, Van Selm JC, Lowenberg M, Ponsioen CY, D'Haens GR, Mathot RA. Explaining Interpatient Variability in Adalimumab Pharmacokinetics in Patients With Crohn's Disease. Ther Drug Monit. 2018 Apr;40(2):202-211. doi: 10.1097/FTD.0000000000000494. PMID 29529008
- [Background] Brandse JF, van den Brink GR, Wildenberg ME, van der Kleij D, Rispens T, Jansen JM, Mathot RA, Ponsioen CY, Lowenberg M, D'Haens GR. Loss of Infliximab Into Feces Is Associated With Lack of Response to Therapy in Patients With Severe Ulcerative Colitis. Gastroenterology. 2015 Aug;149(2):350-5.e2. doi: 10.1053/j.gastro.2015.04.016. Epub 2015 Apr 25. PMID 25917786
- [Background] Brandse JF, Mathot RA, van der Kleij D, Rispens T, Ashruf Y, Jansen JM, Rietdijk S, Lowenberg M, Ponsioen CY, Singh S, van den Brink GR, D'Haens GR. Pharmacokinetic Features and Presence of Antidrug Antibodies Associate With Response to Infliximab Induction Therapy in Patients With Moderate to Severe Ulcerative Colitis. Clin Gastroenterol Hepatol. 2016 Feb;14(2):251-8.e1-2. doi: 10.1016/j.cgh.2015.10.029. Epub 2015 Nov 9. PMID 26545802
- [Background] Brandse JF, Mould D, Smeekes O, Ashruf Y, Kuin S, Strik A, van den Brink GR, D'Haens GR. A Real-life Population Pharmacokinetic Study Reveals Factors Associated with Clearance and Immunogenicity of Infliximab in Inflammatory Bowel Disease. Inflamm Bowel Dis. 2017 Apr;23(4):650-660. doi: 10.1097/MIB.0000000000001043. PMID 28195852
- [Background] Papamichael K, Cheifetz AS. Therapeutic Drug Monitoring in IBD: The New Standard-of-Care for Anti-TNF Therapy. Am J Gastroenterol. 2017 May;112(5):673-676. doi: 10.1038/ajg.2017.21. Epub 2017 Feb 21. No abstract available. PMID 28220781
- [Background] Papamichael K, Vande Casteele N, Ferrante M, Gils A, Cheifetz AS. Therapeutic Drug Monitoring During Induction of Anti-Tumor Necrosis Factor Therapy in Inflammatory Bowel Disease: Defining a Therapeutic Drug Window. Inflamm Bowel Dis. 2017 Sep;23(9):1510-1515. doi: 10.1097/MIB.0000000000001231. PMID 28816757
- [Background] Papamichael K, Baert F, Tops S, Assche GV, Rutgeerts P, Vermeire S, Gils A, Ferrante M. Post-Induction Adalimumab Concentration is Associated with Short-Term Mucosal Healing in Patients with Ulcerative Colitis. J Crohns Colitis. 2017 Jan;11(1):53-59. doi: 10.1093/ecco-jcc/jjw122. Epub 2016 Jul 11. PMID 27402915
- [Background] Seow CH, Newman A, Irwin SP, Steinhart AH, Silverberg MS, Greenberg GR. Trough serum infliximab: a predictive factor of clinical outcome for infliximab treatment in acute ulcerative colitis. Gut. 2010 Jan;59(1):49-54. doi: 10.1136/gut.2009.183095. PMID 19651627
- [Background] Gibson DJ, Heetun ZS, Redmond CE, Nanda KS, Keegan D, Byrne K, Mulcahy HE, Cullen G, Doherty GA. An accelerated infliximab induction regimen reduces the need for early colectomy in patients with acute severe ulcerative colitis. Clin Gastroenterol Hepatol. 2015 Feb;13(2):330-335.e1. doi: 10.1016/j.cgh.2014.07.041. Epub 2014 Jul 30. PMID 25086187
- [Background] Mumolo MG, Bertani L, Ceccarelli L, Laino G, Di Fluri G, Albano E, Tapete G, Costa F. From bench to bedside: Fecal calprotectin in inflammatory bowel diseases clinical setting. World J Gastroenterol. 2018 Sep 7;24(33):3681-3694. doi: 10.3748/wjg.v24.i33.3681. PMID 30197475
- [Background] Rokkas T, Portincasa P, Koutroubakis IE. Fecal calprotectin in assessing inflammatory bowel disease endoscopic activity: a diagnostic accuracy meta-analysis. J Gastrointestin Liver Dis. 2018 Sep;27(3):299-306. doi: 10.15403/jgld.2014.1121.273.pti. PMID 30240474
- [Background] Mosli MH, Zou G, Garg SK, Feagan SG, MacDonald JK, Chande N, Sandborn WJ, Feagan BG. C-Reactive Protein, Fecal Calprotectin, and Stool Lactoferrin for Detection of Endoscopic Activity in Symptomatic Inflammatory Bowel Disease Patients: A Systematic Review and Meta-Analysis. Am J Gastroenterol. 2015 Jun;110(6):802-19; quiz 820. doi: 10.1038/ajg.2015.120. Epub 2015 May 12. PMID 25964225
- [Background] Parente F, Molteni M, Marino B, Colli A, Ardizzone S, Greco S, Sampietro G, Foschi D, Gallus S. Are colonoscopy and bowel ultrasound useful for assessing response to short-term therapy and predicting disease outcome of moderate-to-severe forms of ulcerative colitis?: a prospective study. Am J Gastroenterol. 2010 May;105(5):1150-7. doi: 10.1038/ajg.2009.672. Epub 2009 Dec 8. PMID 19997096
- [Background] Horsthuis K, Bipat S, Bennink RJ, Stoker J. Inflammatory bowel disease diagnosed with US, MR, scintigraphy, and CT: meta-analysis of prospective studies. Radiology. 2008 Apr;247(1):64-79. doi: 10.1148/radiol.2471070611. PMID 18372465
- [Background] Sey MS, Gregor J, Chande N, Ponich T, Bhaduri M, Lum A, Zaleski W, Yan B. Transcutaneous bowel sonography for inflammatory bowel disease is sensitive and specific when performed in a nonexpert low-volume North American center. J Ultrasound Med. 2013 Aug;32(8):1413-7. doi: 10.7863/ultra.32.8.1413. PMID 23887951
- [Background] Yan B, Feagan B, Teriaky A, Mosli M, Mohamed R, Williams G, Yeung E, Yong E, Haig A, Sey M, Stitt L, Zou GY, Jairath V. Reliability of EUS indices to detect inflammation in ulcerative colitis. Gastrointest Endosc. 2017 Dec;86(6):1079-1087. doi: 10.1016/j.gie.2017.07.035. Epub 2017 Jul 29. PMID 28760533
- [Background] Lachin JM. Introduction to sample size determination and power analysis for clinical trials. Control Clin Trials. 1981 Jun;2(2):93-113. doi: 10.1016/0197-2456(81)90001-5. PMID 7273794